CLINICAL TRIAL: NCT00287040
Title: Breast Cancer Screening Via Computer V. Phone
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 0408-03B; R01NR008434 (NIH); NIH: R01 NR0083434
Record Dates: First submitted 2006-02-03; First posted 2006-02-06 (Estimated); Last update posted 2012-05-17 (Estimated); Status verified 2008-08

CONDITIONS: Breast Cancer Screening
Keywords: Breast Cancer; Mammography
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 - Usual Care (No Intervention): This arm looks at mammogram adherence in those individuals who at this time are not receiving booster mammogram interventions.
- 2. DVD Intervention (Experimental): This arm will receive the initial information provided in usual care and will also receive booster mammography interventions via DVD.
  Interventions: Behavioral: Tailored, interactive intervention for mammography screening
- 3. Telephone Counseling (Experimental): This arm will receive the initial information provided in usual care and receive boosters through tailored telephone counseling.
  Interventions: Behavioral: Tailored, interactive intervention for mammography screening

INTERVENTIONS:
Behavioral: Tailored, interactive intervention for mammography screening — Follow ups will occur at 6-, 12-, and 21-months in order to determine effectiveness of intervention as well as cost effectiveness and variation based on participant characteristics to facilitate a more effective program for mammography screenings
  Arms: 2. DVD Intervention; 3. Telephone Counseling

SUMMARY:
The purpose of this study is to compare mammography adherence among women receiving tailored, interactive mammography interventions via DVD and telephone counseling to usual care.

DETAILED DESCRIPTION:
Efficacy Study - We will use stratified block randomization based on race to ensure that the treatment groups maintain comparable race composition. Participants will be randomly assigned to one of the intervention groups or to usual care. Intervention Group 1 will receive, by mail, a DVD version of the interactive computer program; based on responses to its queries, the program will supply immediate feedback to promote mammography. Intervention Group 2 will receive a telephone version of the tailored intervention delivered by a counselor stationed at a computer. The counselor will use questions from the interactive program and deliver messages the program generates in response to each woman's answers. A third group will receive usual care. All women will be asked to participate in 6-month and 21-month follow-up telephone interviews querying stage of mammography adherence and beliefs.

ELIGIBILITY:
Inclusion Criteria:

* • Must have been a member of their HMO/insurance plan for at least 15 months with records indicating no mammogram (screening or diagnostic) in that 15-month period

  * Current member of the plan at time of study enrollment
  * No history of breast cancer diagnosis
  * Complete telephone number and mailing address

Exclusion Criteria:

* • Any claim submitted for a mammogram (screening or diagnostic) in the last 15 months within the HMO/insurance plan or an outside source

  * Previous breast cancer diagnosis
  * Incomplete telephone number or mailing address

Ages: 41 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1686 (Actual)
Dates: Start 2007-09; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
To increase annual mammography adherence | at 6-, 12-, and 21-Months

SECONDARY OUTCOMES:
Cost-effectiveness of DVD versus telephone survey | at 6-, 12-, and 21-months

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Champion, DNS, Principal Investigator — Indiana University
Locations (2):
- United States (2):
  - Indiana University, Indianapolis, Indiana
  - Duke University, Durham, North Carolina

REFERENCES:
- [Derived] Gathirua-Mwangi WG, Monahan PO, Stump T, Rawl SM, Skinner CS, Champion VL. Mammography Adherence in African-American Women: Results of a Randomized Controlled Trial. Ann Behav Med. 2016 Feb;50(1):70-8. doi: 10.1007/s12160-015-9733-0. PMID 26416127
- [Derived] Champion VL, Rawl SM, Bourff SA, Champion KM, Smith LG, Buchanan AH, Fish LJ, Monahan PO, Stump TE, Springston JK, Gathirua-Mwangi WG, Skinner CS. Randomized trial of DVD, telephone, and usual care for increasing mammography adherence. J Health Psychol. 2016 Jun;21(6):916-26. doi: 10.1177/1359105314542817. Epub 2014 Jul 28. PMID 25070967